CLINICAL TRIAL: NCT06913231
Title: Impact of Whole-Body Vibration on Anthropometric Measurement and Body Composition in Overweight and Obese University Students: A Randomized Controlled Trial
Brief Title: Impact of Whole-Body Vibration on Anthropometric Measurement and Body Composition in Overweight and Obese University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rokaia Ali Zainelabedeen Mohamed Toson, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7586
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group (no = 16) underwent whole-body vibration (WBV) training using the PowerPlate device. Sessions will be conducted three times per week for 6 weeks.
  Interventions: Device: Whole body vibration device
- Control group (Sham Comparator): The sham WBV group (no=16) will stand on the same device with the vibtation shut off. Sessions will be conducted three times per week for 6 weeks.
  Interventions: Other: Sham Whole body vibration

INTERVENTIONS:
Device: Whole body vibration device — Whole-body vibration (WBV) training using the Power Plate Pro 7HC (Northbrook, USA). The vibration frequency was set between 30-40 Hz, with an amplitude of 2-4 mm.
  Arms: Study group
Other: Sham Whole body vibration — A sham Whole body vibration will be used . participants will stand on the device without actual vibrations.This control condition will be used to isolate the effects of WBV from other potential influences such as standing posture and time spent on the the platform.
  Arms: Control group

SUMMARY:
Obesity has become a significant public health concern globally, particularly among university students, where lifestyle changes contribute to increased body weight and fat accumulation. The World Health Organization defines obesity as a condition characterized by excessive fat accumulation that presents a risk to health, with a body mass index (BMI) of 30 or higher being a common threshold for classification. In Saudi Arabia, the prevalence of obesity among young adults is alarming, necessitating effective interventions to combat this issue.

ELIGIBILITY:
Inclusion Criteria:

* Male and female University students with BMI ≥ 25, and their age between 18-25 years.

Exclusion Criteria:

* Musculoskeletal, neurological and cardiovacular conditionds,in addition to pregnancy and insrtion of pacemekers or other metal implants.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6 weeks
  BMI will be calculated as weight (kg) divided by height (m²).
Waist circumference | 6 weeks
  WC will be measured at the midpoint between the lower rib and iliac crest using a non-stretchable measuring tape.

SECONDARY OUTCOMES:
Body fat percentage | 6 weeks
  A smart scale will be used to measure body composition including the percentage of whole bofy fat.
Visceral mass | 6 weeks
  Visceral fat will be assesed also using the same smart scale using the bioelectrical impedance analysis.
Lean body mass | 6 weeks
  bioelectrical impedance analysis will be also used via a smart scale to measure the total lean body mass in (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- College of Applied Medical Sciences, Jouf University, Jouf, Sakaka, Saudi Arabia